CLINICAL TRIAL: NCT05655767
Title: Assessment of the pathophysioLogical bAsis of Local Tissue compliaNce Using augmenteD iMAging Techniques to Identify Regional Flow dynamiCs (LANDMARC): a Study With Focus on Aorta Ascendens
Brief Title: LANDMARC Study: a Study With Focus on Aorta Ascendens
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL82141.068.22
Record Dates: First submitted 2022-11-22; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-11

CONDITIONS: Aortic Diseases; Aortic Aneurysm; Aortic Dissection; Aortic Aneurysm, Thoracic; Aortic Dilatation; Aortic Elongation
MeSH Terms: conditions — Aortic Diseases; Aortic Aneurysm; Aortic Dissection; Aortic Aneurysm, Thoracic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 4D-flow MR & CT-scan — 4D-flow MR and CT-scan after cardiac surgery (until 12 months afterwards), for the purpose of obtaining more precise data on (hemo)dynamic processes within the cardiovascular system, in combination with data extraction from the established biobank and databank (FIBAA-bank).

SUMMARY:
Rationale:

Aortic diameter is currently used as a gold standard in international guidelines for prediction of aorta pathology (aortic aneurysm and aortic dissection). However, aortic diameter has proven to be insufficiently accurate for making decisions about well-timed preventive interventions. The LANDMARC study will take place in line with the FIBAA-bank ('Correlatie tussen cardiovasculaire FIBroseringsgraad en Aorta elongatie, dilatatie en Atria dilatatie (FIBAA-bank): een biobank & databank onderzoek met focus op aorta en atria' (METC-number 2022-3164)), and aims to reveal the undiscovered relationship between WSS (wall shear stress) values and aortic strain. In combination with data from the FIBAA-bank, the LANDMARC study will provide more accurate information for future risk stratification models for cardiovascular pathology (with focus on aortic disease).

Objectives:

Primary objective: indication of the association between WSS (peak WSS and WSS gradient) (through 4D-flow MR and CT) and aortic strain.

Secondary objective: indication of the association between (hemo)dynamic processes within the body (aortic elongation/aortic strain) and (patho-)physiological changes (degree of cardiovascular tissue fibrosis).

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Able to understand the trial and provide informed consent
* Patients who have participated in the FIBAA-bank

Exclusion Criteria:

* Patients with abnormal congenital cardiothoracic anatomy, with exception of presence of a bicuspid aortic valve
* Patients with history of chemotherapy, or radiotherapy within thoracic region
* Patients with an age >80 years
* Patients with a weight >120 kg
* Patients with a contra-indication for MRI according to the MUMC+ ODIN protocol nr. 004952
* Patients with impaired renal function (GFR <30)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population of the LANDMARC study will consist of patients who underwent open heart surgery and have participated in FIBAA-bank.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2022-12-15 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Indication of the association between WSS (peak WSS and WSS gradient) (through 4D-flow MR and CT) and aortic strain. | Until 12 months postoperative
  Previous research described the importance of aortic strain for the prediction of aortic disease. By linking this information to information that can be obtained via advanced imaging techniques, future predictions about aortic disease can be made more easily and will be more accurate.

SECONDARY OUTCOMES:
Indication of the association between (hemo)dynamic processes within the body (aortic elongation/aortic strain) and (patho-)physiological changes (degree of cardiovascular tissue fibrosis). | Until 12 months postoperative
  During the FIBAA bank, residual tissue (e.g. aorta and atrial tissue) and blood (25ml) were collected, which were then analysed by the Biochemistry department. From these materials, data on for example elasticity and compliance was collected using different staining techniques (elastin-collagen ratio, type I-type II collagen ratio, degree of collagen fibre crosslinking, etc.). This available data is used during the LANDMARC study to indicate associations between degree of cardiovascular tissue fibrosis and aortic elongation/aortic strain.
  These associations will demonstrate that cardiovascular tissue response and cell interaction based on dynamic body processes and hemodynamics are important factors for the development of cardiovascular disease.

CONTACTS AND LOCATIONS:
Locations (1):
- MaastrichtUMC, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided